CLINICAL TRIAL: NCT07061951
Title: A Phase 2 Pilot Study of Mirdametinib in Relapsed Refractory Chronic Lymphocytic Leukemia
Brief Title: Testing the Effectiveness of the Anti-cancer Drug, Mirdametinib, in Treating Relapsed, Refractory Chronic Lymphocytic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-04637; NCI-2025-04637 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10708 (Other: Dana-Farber - Harvard Cancer Center LAO); 10708 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2025-07-11; First posted 2025-07-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Specimen Handling; Biopsy; mirdametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (mirdametinib) (Experimental): Patients receive mirdametinib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo bone marrow biopsy, blood sample collection, echocardiography, and CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Mirdametinib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Drug: Mirdametinib — Given PO
  Other Names: Gomekli; MEK Inhibitor PD0325901; PD 901; PD-0325901

SUMMARY:
This phase II trial tests the effect of mirdametinib in treating patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). Mirdametinib, a methyl ethyl ketone (MEK) inhibitor, works by blocking the action of an abnormal protein that signals cancer cells to multiply. This may help slow or stop the spread of cancer cells. Giving mirdametinib may be effective in treating patients with relapsed or refractory CLL or SLL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the best objective response rate (ORR) with single agent mirdametinib. ORR will be composed of complete response (CR), CR with incomplete marrow recovery (CRi), and partial remission (PR) as defined by the 2018 Modified International Workshop on Chronic Lymphocytic Leukemia (iwCLL) National Cancer Institute-Working Group (NCI-WG) criteria, which includes PR with lymphocytosis (Hallek et al., 2018).

SECONDARY OBJECTIVES:

I. To determine the effect of mirdametinib on progression-free survival (PFS). II. To evaluate the duration of response (DOR) for mirdametinib in relapsed refractory chronic lymphocytic leukemia (R/R CLL).

III. To determine the effect of mirdametinib on overall survival (OS). IV. To evaluate the safety and tolerability of mirdametinib, including the rates of high grade (3+) events, and rates of discontinuations and dose modifications.

OUTLINE:

Patients receive mirdametinib orally (PO) twice daily (BID) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo bone marrow biopsy, blood sample collection, echocardiography, and computed tomography (CT) throughout the study.

After completion of study treatment, patients are followed up at 30 days then every 2 months until starting a new therapy followed by every 3 months for up to a total of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed CLL or small lymphocytic lymphoma (SLL), as documented by a history at some point in time of an absolute peripheral blood B cell count > 5000/mcL with a monoclonal B cell population coexpressing CD19, CD5, and CD23, or if CD23 negative, then documentation of the absence of t(11;14) or cyclin D1 overexpression. Alternatively, patients with lymphadenopathy in the absence of circulating disease will also be eligible for this study if lymph node biopsy or bone marrow biopsy has established the diagnosis of CLL with the above immunophenotype
* Patients must have a current indication for treatment as defined by the iwCLL 2018 Guidelines (Hallek et al., 2018):

  * Massive or progressive splenomegaly; OR
  * Massive lymph nodes, nodal clusters, or progressive lymphadenopathy; OR
  * Grade 2 or 3 fatigue; OR
  * Fever ≥ 100.5°F or night sweats for greater than 2 weeks without documented infection; OR
  * Presence of weight loss ≥ 10% over the preceding 6 months; OR
  * Progressive lymphocytosis with an increase of ≥ 50% over a 2-month period or an anticipated doubling time of less than 6 months; OR
  * Evidence of progressive marrow failure as manifested by the development of or worsening of anemia and or thrombocytopenia
* Patients must have measurable disease, defined as lymphocytosis > 5,000/mcL, palpable or computed tomography (CT) measurable lymphadenopathy > 1.5 cm, or bone marrow involvement > 30%
* Patients must have received at least two prior therapies for CLL including systemic therapy containing a Bruton's tyrosine kinase (BTK) inhibitor and a BCL2 inhibitor. Patients are required to have prior BTK inhibitor-based therapy because constitutive extracellular signal-regulated kinase (ERK) activation is seen in all patients with progression after BTK inhibitor therapy
* Age ≥ 18 years. Because CLL is extremely rare in persons < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Absolute neutrophil count ≥ 500/mcL. Growth factor is allowed to achieve this level. Neutrophil count of 250 is permitted for patients with bone marrow involvement

  * Unless they have significant bone marrow involvement of CLL confirmed on biopsy
* Platelets ≥ 20,000/mcL independent of transfusion within 7 days of screening. Transfusion is permitted to support platelet count for patients with bone marrow involvement

  * Unless they have significant bone marrow involvement of CLL confirmed on biopsy
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) unless bilirubin rise is due to Gilbert's syndrome, autoimmune hemolytic anemia,(AIHA), or of non-hepatic origin
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x institutional ULN
* Glomerular filtration rate (GFR) 50 ml/min estimated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) (Levey et al., 2009)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* The effects of mirdametinib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use highly effective contraception (hormonal and barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women of child-bearing potential should also use adequate contraception for 6 months after completion of mirdametinib administration. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of mirdametinib administration. Women of childbearing age should not donate egg(s) and men should not donate sperm for the duration of study participation and 3 months after completion of mirdametinib administration

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to mirdametinib
* Patients with concurrent administration of strong inhibitors and inducers of P-glycoprotein (P-g)p or breast cancer specific resistance protein (BCRP). If discontinuation of the medication is appropriate, a washout duration of approximately 3 to 5 half-lives is recommended prior to the first dose of mirdametinib
* Patients with concurrent administration of strong CYP3A4 inducers. If discontinuation of the medication is appropriate, a washout duration of approximately 3 to 5 half-lives is recommended prior to the first dose of mirdametinib
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant women are excluded from this study because mirdametinib is MEK inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother mirdametinib, breastfeeding should be discontinued if the mother is treated with mirdametinib
* Patients with active infection requiring intravenous (IV) antibiotics
* History or current evidence of glaucoma or clinically significant abnormalities on the ophthalmological exam, including but not limited to cataract limiting the ability to examine the retina or any optical coherence tomography (OCT) finding that could be a significant risk factor for retinal vein occlusion (RVO), retinopathy, or neovascular macular degeneration
* Patients with corrected QT (QTc) > 470 ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-09-08 (Estimated); Primary Completion 2030-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Best objective response rate | Up to 5 years
  Will be defined as the best achieved response (e.g., complete response [CR], CR with incomplete marrow recovery, partial remission [PR], PR with lymphocytosis) as determined by International Workshop on Chronic Lymphocytic Leukemia criteria. Will be summarized descriptively.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 5 years
  The Kaplan Meier method will be used to estimate the median PFS time and PFS.
Duration of response | Up to 5 years
  Will be summarized descriptively.
Overall survival | Up to 5 years
Incidence of adverse events (AEs) | Up to 30 days after last dose of study treatment
  Will be described and graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.
Incidence of high grade (3+) AEs | Up to 30 days after last dose of study treatment
  Will be described and graded using NCI CTCAE v 5.0.
Rates of discontinuation and dose interruptions | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R Brown, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (1):
- Dana-Farber - Harvard Cancer Center LAO, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm